CLINICAL TRIAL: NCT00960076
Title: 18-Week, Multicenter, Randomized, Double-Blind 3b Trial to Evaluate Efficacy/Safety of Saxagliptin in Combo With Metformin XR 1500mg vs Metformin Uptitrated to 2000mg in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control After Diet/Exercise and a Stable Dose of Metformin XR 1500mg
Brief Title: An 18 Week Efficacy and Safety Study of Saxagliptin and Metformin XR Combination in Subjects With Type 2 Diabetes
Acronym: SCORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1680L00005
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Results first posted 2011-09-27 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes
Keywords: T2DM; Metformin; A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Saxagliptin
  Interventions: Drug: Saxagliptin; Drug: Metformin XR
- 2 (Active Comparator): Metformin Extended Release
  Interventions: Drug: Metformin XR

INTERVENTIONS:
Drug: Saxagliptin — 5mg oral tablet once daily
  Other Names: Onglyza
  Arms: 1
Drug: Metformin XR — 500mg oral tablet once daily
  Arms: 2
Drug: Metformin XR — 750mg, 2 tablets once daily

SUMMARY:
The purpose of this study is to compare reduction in A1C for subjects taking Saxagliptin and Metformin XR vs. uptitrated Metformin XR.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetics taking metformin IR or XR greater than or equal to 850mg and less than or equal to 1500mg only for at least 8 weeks prior to screening
* A1c: 7.5-11% (at screening)
* BMI less than or equal to 45 kg/m2

Exclusion Criteria:

* Significant cardiovascular history
* Active liver disease, renal impairment

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boaz Hirschberg, MD, Study Director — AstraZeneca; Vivian Fonseca, MD, Principal Investigator — Tulane University
Locations (35):
- United States (22):
  - Research Site, Jonesboro, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Fountain Valley, California
  - Research Site, Los Angeles, California
  - Research Site, Pasadena, California
  - Research Site, Sacramento, California
  - Research Site, Gainesville, Florida
  - Research Site, Wellington, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, St Louis, Missouri
  - Research Site, Salisbury, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Simpsonville, South Carolina
  - Research Site, Bristol, Tennessee
  - Research Site, Alexandria, Virginia
  - Research Site, Burke, Virginia
  - Research Site, Manassas, Virginia
- Colombia (3):
  - Research Site, Barranquilla, Atlántico
  - Research Site, Barranquilla
  - Research Site, Bogotá
- Costa Rica (3):
  - Research Site, Curridabat, Provincia de San José
  - Research Site, Los Yoses, Provincia de San José
  - Research Site, Heredia
- Mexico (6):
  - Research Site, México, D.f.
  - Research Site, Durango, Durango
  - Research Site, Guadalajara, Jalisco
  - Research Site, Zapopan, Jalisco
  - Research Site, Cuernavaca, Morelos
  - Research Site, Querétaro City, Querétaro
- Research Site, Lima, Peru

REFERENCES:
- [Derived] Fonseca V, Zhu T, Karyekar C, Hirshberg B. Adding saxagliptin to extended-release metformin vs. uptitrating metformin dosage. Diabetes Obes Metab. 2012 Apr;14(4):365-71. doi: 10.1111/j.1463-1326.2011.01553.x. Epub 2012 Jan 18. PMID 22192246

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 393 subjects who entered the lead-in period, 111 subjects did not enter the randomized, double-blind treatment period. Thus, a total of 282 subjects were randomized and treated.
Groups:
- Saxagliptin + Metformin: Saxagliptin 5 mg (DB) + Metformin XR 1500 mg (OL)
- Metformin (DB) + Metformin (OL): Metformin XR 500 mg (DB) + Metformin XR 1500 mg (OL)
Period: Overall Study
Arm/Group | Saxagliptin + Metformin | Metformin (DB) + Metformin (OL)
Started | 138 (Randomized and treated) | 144 (Randomized and treated)
Completed | 130 (Completing 18 weeks of treatment) | 119 (Completing 18 weeks of treatment)
Not Completed | 8 | 25
Not completed — Adverse Event | 1 | 7
Not completed — No longer met study criteria | 1 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 3 | 3
Not completed — Severe non-compliance to protocol | 1 | 2
Not completed — Hyperglycemia | 1 | 5
Not completed — Did not attend the termination visit | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin + Metformin | Metformin (DB) + Metformin (OL) | Total
Number analyzed (Participants) | 138 | 144 | 282
Age Continuous [Mean (Standard Deviation); unit: years] | 55.22 (9.41) | 55.46 (9.86) | 55.34 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 71 | 152
  Male | 57 | 73 | 130

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c Level From Baseline to Week 18 (LOCF)
Description: Adjusted mean change from baseline in HbA1c achieved with saxagliptin added on to metformin versus metformin at Week 18 (Randomized Analysis Set). HbA1c is a continuous measure, the change from baseline for each participant is calculated as the Week 18 value minus the baseline value.
Time Frame: Baseline to week 18
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Saxagliptin + Metformin | Metformin (DB) + Metformin (OL)
Number analyzed (Participants) | 137 | 142
Percent
  Baseline | 8.41 (0.076) | 8.28 (0.077)
  Week 18 | 7.53 (0.093) | 7.93 (0.111)
  Adjusted Change from Baseline to Week 18 | -0.88 (0.077) | -0.35 (0.076)
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Metformin (DB) + Metformin (OL); Test type: Superiority or Other; Mean Difference (Net) = -0.52, 95% CI 2-sided [-0.73 to -0.31], Standard Error of Mean 0.108

2. Secondary Outcome: Change in 2-hour PPG Following Mixed Meal Tolerance Test (MMTT) From Baseline to Week 18 (LOCF)
Description: Adjusted mean change from baseline in 2-hour PPG (following MMTT) achieved with saxagliptin added on to metformin versus metformin at Week 18 (Randomized Analysis Set). PPG is a continuous measure, the change from baseline for each participant is calculated as the Week 18 value minus the baseline value.
Time Frame: Baseline to week 18
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin + Metformin | Metformin (DB) + Metformin (OL)
Number analyzed (Participants) | 121 | 117
mg/dL
  Baseline | 227.36 (6.022) | 223.68 (5.295)
  Week 18 | 195.11 (5.876) | 216.24 (6.230)
  Adjusted Change from Baseline to Week 18 | -31.52 (4.996) | -8.20 (5.081)
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Metformin (DB) + Metformin (OL); Test type: Superiority or Other; Mean Difference (Net) = -23.32, 95% CI 2-sided [-37.36 to -9.28], Standard Error of Mean 7.128

3. Secondary Outcome: Change in FPG From Baseline to Week 18 (LOCF)
Description: Adjusted mean change from baseline in FPG achieved with saxagliptin added on to metformin versus metformin at Week 18 (Randomized Analysis Set). FPG is a continuous measure, the change from baseline for each participant is calculated as the Week 18 value minus the baseline value.
Time Frame: Baseline to week 18
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin + Metformin | Metformin (DB) + Metformin (OL)
Number analyzed (Participants) | 137 | 142
mg/dL
  Baseline | 162.54 (4.146) | 163.35 (3.910)
  Week 18 | 142.70 (3.633) | 156.32 (3.948)
  Adjusted Change from Baseline to Week 18 | -20.03 (3.146) | -6.85 (3.090)
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Metformin (DB) + Metformin (OL); Test type: Superiority or Other; Mean Difference (Net) = -13.18, 95% CI 2-sided [-21.86 to -4.50], Standard Error of Mean 4.409

4. Secondary Outcome: Percent of Subjects Reaching Goal (HbA1c <7%) at Week 18 (LOCF) - Percent of Subjects (1)
Description: Percent of subjects achieving therapeutic response (HbA1c <7.0%) at Week 18 (LOCF) (Randomized analysis set)
Time Frame: Week 18 (LOCF)
Measure: Number; unit: Percentage of Participants
Arm/Group | Saxagliptin + Metformin | Metformin (DB) + Metformin (OL)
Number analyzed (Participants) | 137 | 142
Percentage of Participants | 37.2 | 26.1
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Metformin (DB) + Metformin (OL); Test type: Superiority or Other; p = 0.0459, ANCOVA; Mean Difference (Net) = 11.2, 95% CI 2-sided [0.2 to 22.0]

ADVERSE EVENTS:
Arm/Group | Saxagliptin + Metformin | Metformin (DB) + Metformin (OL)
Serious Adverse Events (participants affected / at risk) | 0/138 | 3/144
Other Adverse Events (participants affected / at risk) | 21/138 | 16/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin + Metformin (N=138) | Metformin (DB) + Metformin (OL) (N=144)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin + Metformin (N=138) | Metformin (DB) + Metformin (OL) (N=144)
Urinary Tract Infection (Infections and infestations) | 7 | 3
Nasopharyngitis (Infections and infestations) | 6 | 8
Diarrhoea (Gastrointestinal disorders) | 8 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No